CLINICAL TRIAL: NCT02828852
Title: Study of the Platelet Function During the Last Month of Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 09 163 02; Local Grant 2009 (Other Grant/Funding Number: 0916302)
Record Dates: First submitted 2016-07-04; First posted 2016-07-12 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Pregnancy
Keywords: pregnancy; platelets
MeSH Terms: interventions — Blood Specimen Collection; Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pregnancy (Experimental): Blood sample
  Interventions: Other: Blood sample
- No pregnancy (Experimental): Blood sample
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — In washed platelets and whole blood, study shall determine the percentage of aggregation after activation by different agonists and the amount of certain membrane markers of platelet activation. Furthermore, an assay of estradiol plasma will be made.
  In whole blood, study will evaluate the percentage of platelet adhesion to collagen matrix or fibrinogen and the volume of thrombies formed.
  Other Names: Blood sample in pregnancy and no pregnancy women

SUMMARY:
The objective is to compare women's platelet answer in the last month of pregnancy to women old enough to procreate, no pregnancy and without hormonal treatment.

The hypothesis of research is that the decrease of platelet answer in pregnant women could not only limit the occurence of embolic accidents but also explain the lowest incidence of the arterial thrombosis in comparison with the venous thrombosis.

DETAILED DESCRIPTION:
This is a monocentric study comparing a group of pregnant women and a group of "no pregnancy" women.

The goal of the present study is to determine the impact of pregnancy on platelet function. For this, the study propose to explore, in women in the last month of pregnancy, the ability of platelets to aggregate after activation by strong agonists but also their ability to adhere to a matrix and form thrombies.

The study will include 30 pregnant and 30 "no pregnancy" control women, of childbearing age and not taking hormone therapy. From a blood sample, two types of examination will be implemented:

A) In whole blood, we will evaluate the percentage of platelet adhesion to collagen matrix or fibrinogen and the volume of thrombies formed.

B) In washed platelets and whole blood, we shall determine the percentage of aggregation after activation by different agonists and the amount of certain membrane markers of platelet activation. Furthermore, an assay of estradiol plasma will be made.

ELIGIBILITY:
Inclusion Criteria:

* Signature of the form of consent
* Absence of any physical or psychic pathology which can interfere with the normal realization of the study

  * Group1 : Women in the last month of pregnancy
  * Group 2 : Women old enough to procreate, no pregnancy and without hormonal treatment

Exclusion Criteria:

* Thrombopenia (platelet numeration < 120 000 / mm3),
* Gestational diabet,
* Hormonal treatment : oestrogen-progestagen, progestagen, Selective Estrogen Receptor Modulator (SERM), inductors of ovulation,
* Anticoagulant and any medication which can intervene on the platelet function (AINS, antidepressants)
* Personal history of thromboembolic accident venous or arterial,
* Personal history of haemostasis disease
* Personal history of hepatic or renal disease
* Personal history of autoimmune disease.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2010-05; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
surface covered by platelets | baseline
  Percentage of surface covered by platelets (using the software Metamorph)
Volume of thrombies | baseline
  Total volume of thrombies in μm3 (using the software Metamorph)

SECONDARY OUTCOMES:
Platelet aggregation | baseline
  Percentage of platelet aggregation (whole blood and washed platelets)
chemokine Platelet Factor 4 | baseline
  Quantity of the chemokine Platelet Factor 4 (PF4) (IU/ml) secreted by the granules after activation by these agonists (washed platelets)
Thromboglobulin | baseline
  Quantity of thromboglobulin (in ng / ml) secreted by the granules after activation by these agonists (washed platelets)

CONTACTS AND LOCATIONS:
Overall Officials: PARANT Olivier, MD PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital of Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Valera MC, Parant O, Cenac C, Arnaud C, Gallini A, Hamdi S, Sie P, Arnal JF, Payrastre B. Platelet Adhesion and Thrombus Formation in Whole Blood at Arterial Shear Rate at the End of Pregnancy. Am J Reprod Immunol. 2015 Dec;74(6):533-41. doi: 10.1111/aji.12433. Epub 2015 Oct 4. PMID 26435170